CLINICAL TRIAL: NCT01391078
Title: Comparison of Sensimed Triggerfish (TF) 24 Hour IOP Monitoring With Goldmann Applanation Tonometry (GAT) and Perkins Tonometry in Glaucoma Patients
Brief Title: Comparison of Sensimed Triggerfish With Goldmann Applanation Tonometry and Perkins Tonometry
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Katrin Lorenz (Other)
Collaborators: Sensimed AG (Industry)
Responsible Party: Sponsor-Investigator, Katrin Lorenz, MD, Johannes Gutenberg University Mainz
Organization: Johannes Gutenberg University Mainz (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: Sensimed Triggerfish11/01
Record Dates: First submitted 2011-06-14; First posted 2011-07-11 (Estimated); Last update posted 2012-11-28 (Estimated); Status verified 2012-11

CONDITIONS: Primary Open Angle Glaucoma
Keywords: glaucoma; IOP; Sensimed Triggerfish; Goldmann Applanation Tonometry; fluctuation; comparison
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sensimed Triggerfish (Experimental)
  Interventions: Device: Sensimed Triggerfish Sensor
- Goldmann Applanation Tonometry/Perkins Tonometry (Active Comparator)
  Interventions: Device: Goldmann Applanation Tonometry, Perkins Tonometry

INTERVENTIONS:
Device: Sensimed Triggerfish Sensor — IOP will be monitored for 24 hours
  Arms: Sensimed Triggerfish
Device: Goldmann Applanation Tonometry, Perkins Tonometry — IOP will be measured every two hours within 24 hours
  Arms: Goldmann Applanation Tonometry/Perkins Tonometry

SUMMARY:
This prospective, crossover study is designed to correlate SENSIMED Triggerfish® (TF) continuous IOP monitoring with conventional 24 h intraocular pressure profiles in glaucoma patients. There are two control measurements: The GAT/Perkins profile in the same eye in the second night and the GAT/Perkins profile in the same night in the fellow eye. Therefore, each eye serves as test eye and also as control for the second test eye.

ELIGIBILITY:
Inclusion Criteria:

* Patient is able to comply with the study procedure
* Patient must be ≥ 18 years old
* Diagnosis of primary open angle glaucoma (EGS criteria)
* Similar behaviour of IOP in both eyes in former IOP profiles
* Patient has consented to be in the trial and signed informed consent is available before any study related procedures are carried out
* Visual Acuity of 20/200 or better in both eyes
* Ability of subject to understand the character and individual consequences of the study
* For women with childbearing potential, adequate contraception

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-06; Primary Completion 2012-01 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Relation of GAT/Perkins with TF in a cross-over regression analysis. | 48 hours
  Correlation of GAT/Perkins values with TF data (mean, min, max, fluctuation)

SECONDARY OUTCOMES:
Correlation of IOP in the test eye (TF) compared to a conventional 24h IOP profile (GAT) the reference eye (same night) | 48 hours
  Correlation of GAT/Perkins values with TF data (mean, min, max, fluctuation)
Correlation of IOP profile (GAT) right versus left eye | 48 hours
  Correlation of GAT/Perkins values in the right and left eye (mean, min, max, fluctuation)
Correlation of IOP profile (TF) right versus left eye | 48 hours
  Correlation of TF data right and left eye (mean, min, max, fluctuation)
Correlation of IOP with blood pressure | 48 hours
  Correlation of GAT/Perkins values and TF data with systolic and diastolic blood pressure(mean, min, max, fluctuation)
Correlation of IOP with heart rate | 48 hours
  Correlation of GAT/Perkins values and TF data with pulse rate(mean, min, max, fluctuation)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Ophthalmology, University Medical Center, Johannes Gutenberg-University Mainz, Mainz, RLP, Germany